CLINICAL TRIAL: NCT04576169
Title: TREatment of Triangular FibrOcaRtilage ComplEx Ruptures (REINFORCER): Protocol for Randomized, Controlled, Blinded, Efficacy Trial of Triangular Fibrocartilage Complex Tears
Brief Title: Trial Comparing Treatment Strategies in Triangular Fibrocartilage Complex Ruptures
Acronym: REINFORCER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Kuopio University Hospital (Other); Oulu University Hospital (Other); Karolinska Institutet (Other); Hospital Sønderjylland (Unknown); Copenhagen University Hospital at Herlev (Other); Hospital Nova of Central Finland (Unknown)
Responsible Party: Principal Investigator, Jarkko Jokihaara, Associate professor of hand surgery, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tampere University Hospital
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Triangular Fibrocartilage Complex Injury
Keywords: Arthroscopy; Surgery; Triangular Fibrocartilage; Randomized Controlled Trial; Placebo; Repair; Wrist; Debridement
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Operating surgeon, operating theatre staff, coordinating research assistant (CRA), and research assistants (RA) cannot be blinded to the allocation. In central or radial tear randomization cohort, outcome assessors will be blinded and they will not participate in the care at any other point in the trial, except during follow-up visits. The participants are also blinded, resulting in a triple-blinded randomization cohort since also trialist are blinded in data analysis phase as in foveal tear randomization cohort. In the ulnar tear cohort, randomization cannot be blinded due to differing postoperative treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Central or Radial Tear: Arthroscopic debridement (Experimental): Arthroscopic debridement
  Interventions: Procedure: Arthroscopic Debridement
- Central or Radial Tear: Sham surgery (Placebo Comparator): Diagnostic arthroscopy only (placebo surgery).
  Interventions: Procedure: Placebo surgery
- Ulnar Tear: Arthroscopic or open repair (Experimental): Arthroscopic or open repair
  Interventions: Procedure: Arthroscopic or Open Repair
- Ulnar Tear: Physiotherapy (Active Comparator): Diagnostic arthroscopy and physiotherapy
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Arthroscopic Debridement — Wrist arthroscopy can be performed with or without irrigation. In the debridement arm, a central or radial TFCC tear found during arthroscopy is debrided with a shaver. Portals are closed either with sutures or with medical tape. Immediate mobilization of the wrist is allowed after the operation. Participants are provided with instructions for home exercises, and they are advised to commence the exercises two weeks post-operation.
  Arms: Central or Radial Tear: Arthroscopic debridement
Procedure: Placebo surgery — Diagnostic wrist arthroscopy can be performed with or without irrigation. A central or radial TFCC tear found during wrist arthroscopy is left untouched and no other operative interventions are done. Portals are closed either with sutures or with medical tape. The procedure is performed in general or regional anesthesia in operating room. Participants are not able to see to the operation area or monitor. They will listen to music with noise-cancelling headphones throughout the operation. The operative time will be matched, with the surgeon simulating a debridement procedure. Immediate mobilization of the wrist is allowed after the operation. Participants are provided with instructions for home exercises, and they are advised to commence the exercises two weeks post-operation.
  Arms: Central or Radial Tear: Sham surgery
Procedure: Arthroscopic or Open Repair — An ulnar TFCC tear found during wrist arthroscopy is sutured to the capsule or fovea with one of the separately defined methods choosed by the treating hand surgeon. The procedure is performed in general or regional anesthesia in operating room. Wounds are closed and standardized post-operative treatment is started after six weeks.
  Arms: Ulnar Tear: Arthroscopic or open repair
Procedure: Physiotherapy — An ulnar TFCC tear found during wrist arthroscopy is left untouched and no other operative interventions are done. Portals are closed with sutures or medical tape. The procedure is performed in general or regional anesthesia in operating room. Physiotherapy exercises of wrist and DRUJ stabilizers is started after two weeks.
  Arms: Ulnar Tear: Physiotherapy

SUMMARY:
The trial is a multicentre, randomized, superiority, controlled, participant and outcome assessor (debridement versus placebo surgery randomization cohort) and trialist blinded (both arms) superiority, umbrella trial with two randomized cohorts (1. debridement or placebo surgery, 2. repair or physiotherapy) which both include two 1:1 parallel arms. The primary objective is to investigate the superiority of 1) debridement over placebo surgery and 2) repair over physiotherapy in two randomized cohorts using Patient-Rated Wrist Evaluation (PRWE) at one year post randomisation as the primary outcome.

DETAILED DESCRIPTION:
Triangular fibrocartilage complex (TFCC) injuries are often considered the cause of ulnar wrist pain. TFCC lesions can be traumatic or degenerative according to classification suggested by Palmer and Atzei. Primary treatment is conservative, but if symptoms persist, operative treatment is an option. Depending on the morphology of the tear, the treatment can be either debridement or repair. Trialists have observed improvement of symptoms after TFCC repair but all these trials are observational cohorts without proper controls. Efficacy of surgery has not been studied in randomized controlled trial (RCT) setting.

The investigators planned a multicentre, randomized, superiority, controlled, participant and outcome assessor (debridement versus placebo surgery randomisation cohort) and trialist blinded (both arms) superiority, umbrella trial with two randomized cohorts which both include two 1:1 parallel arms. Participants in the first cohort (central or radial TFCC tear) will undergo randomization to either arthroscopic debridement or placebo surgery. In the second cohort (peripheral TFCC tear), participants will be randomized to arthroscopic/open TFCC repair or physiotherapy. Our primary objective is to investigate the superiority of 1) debridement over placebo surgery for central (Palmer 1A) and radial (Palmer 1D) TFCC tears, and 2) repair over non-operative treatment (physiotherapy) for ulnar (Palmer 1B) TFCC tears in two randomized cohorts using Patient-Rated Wrist Evaluation (PRWE) at one year post randomisation as the primary outcome.

Institutional Review Board (IRB) of Tampere university hospital has approved the study protocol. All participants will give written informed consent. The results of the trial will be disseminated as published articles in peer-reviewed journals.

Outcome measures for different studies are often derived from what clinicians, rather than patients, thinks to be important. The investigators chose to base the efficacy assessment on the measure of patient's subjective disability and pain.

There is no clear evidence of the efficacy of the treatments (debridement and repair). It is justified and ethically correct to compare these treatments to placebo surgery and physiotherapy. Placebo surgery and physiotherapy are less invasive than debridement and repair and because of this are even safer to patients than comparable treatments.

ELIGIBILITY:
Inclusion Criteria:

* Ulnar sided wrist pain
* Age more than 18 years
* Suspicion of TFCC tear in clinical examination
* Ability to fill the Danish, Finnish or Swedish versions of questionnaires
* Symptom duration more than 3 months, and unsuccessful non-operative treatment
* Central (Palmer 1A), ulnar (Palmer 1B) or radial (Palmer 1D) TFCC tear explaining the pain in arthroscopy

Exclusion Criteria:

* Gross instability of DRUJ which will be defined as "obvious instability in clinical examination in each forearm and wrist position"
* Distal (Palmer 1C) TFCC tear in arthroscopy
* Ulnocarpal or DRUJ arthrosis (Atzei class 5)
* Ulnar variance ≥ +2 mm in x-ray
* Age above 65 years
* Rheumatoid arthritis or other inflammatory disease effecting radio- or ulnocarpal or DRUJ
* Lunotriquetral instability diagnosed in arthroscopy
* ECU instability
* Massive tear and degenerated edges or frayed tear which fails suture (Atzei class 4A-4B)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2035-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Wrist Evaluation (PRWE) | 10 year follow-up, primary time point at 1 year
  The PRWE questionnaire is a wrist-specific instrument comprising a 15-item questionnaire assessing pain and disability in daily living. PRWE provides a score ranging from 0 (best) to 100 (worst). This wrist-specific tool demonstrates good reliability, validity, and responsiveness. Translation and validation have been conducted for Danish, Finnish, and Swedish languages. In interpreting the results, we will employ the Minimally Important Difference (MID) value of 14. PRWE as secondary outcome will be measured at all the other time points (6 months, 2, 5 and 10 years) than primary outcome.

SECONDARY OUTCOMES:
Quality of life (EQ-5D-3L) | 10 year follow-up
  The EQ-5D-3L is a widely employed, health-related quality of life instrument comprising five dimensions and a visual VAS for health level. The five dimensions assessed by EQ-5D-3L include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, patients rate their current state on each dimension using a 3-point scale, and the VAS scale ranges from 0 (worst) to 100 (best). Utility or preference weights, applied with an aggregation formula, yield a single index number used to evaluate overall health-related quality of life. It has been proven to be a reliable and validated tool and it is widely used in healthcare research. The EQ-5D-3L has demonstrated good responsiveness in upper extremity conditions, such as distal radius fractures, its responsiveness in hand surgery has not been measured previously. The MID for the index is 0.085 and for the VAS 6.41. Translation and validation for Danish, Finnish, and Swedish languages have been conducted.
Adverse and serious adverse events | 10 year follow-up
  All wrist-related adverse events will be documented: ligament, nerve, tendon, or vascular injury; fracture; CRPS; infection; chondral lesion; hematoma; or any other condition that can be attributed to the intervention. Participants are instructed to promptly notify the outpatient clinic at their center if they detect a potential adverse event. Additionally, adverse events will be assessed during each follow-up visit. Any events resulting in hospitalization or death will be classified as SAE.
Global improvement | 10 year follow-up
  Patient-rated global improvement will be assessed using the question: "How would you rate the function and pain of your wrist compared to the situation before the treatment?" Participants will provide responses on a 7-step Likert scale, ranging from "Much worse" to "Much better.". This global rating of the treatment effect offers a subjective evaluation of the participant's perception of the treatment's impact on their wrist condition. It enables participants to offer feedback on their overall experience and evaluate the practical significance of the treatment's effect on their wrist. The Likert scale, a simple and effective tool for assessing participant-evaluated global ratings, is widely used in clinical research.
Pain in activity | 10 year follow-up
  Pain during activity will be evaluated using the VAS, a validated and reliable tool for pain assessment. Widely employed in pain assessments, the VAS scale ranges from 0 to 100 mm, with higher values indicating more severe pain. The MID for VAS-pain is reported to fall between 16-19 mm.
Grip strength | 2 year follow-up
  Grip strength will be assessed using the Jamar dynamometer, known for its good within-instrument reliability (Spearman Rho correlation coefficient test 0.82). The strength measurement will be performed with the handle in two positions: with the elbow in 90° flexion and the arm in adduction. Results will be reported in kilograms. The MID of grip strength is reported to be 5.5 kg.
ROM of forearm and wrist | 2 year follow-up
  Passive ROM of the forearm and wrist are commonly employed as outcomes in studies addressing the treatment of wrist pathologies. Prosupination, recorded as forearm ROM, will be measured with the elbow at 90° flexion. Wrist ROM measurements will include extension, flexion, ulnar deviation, and radial deviation. MID of forearm and wrist ROM have not been determined.

CONTACTS AND LOCATIONS:
Overall Officials: Antti Kaivorinne, M.D., Principal Investigator — Tampere University Hospital; Mikko P Räisänen, M.D., Principal Investigator — Tampere University Hospital; Teemu Karjalainen, M.D., Ph.D., Principal Investigator — Hospital Nova of Central Finland; Aleksi Reito, M.D., Ph.D., Adjunct professor, Principal Investigator — Tampere University Hospital; Robert Gvozdenovic, M.D., Ph. D., Principal Investigator — Copenhagen University Hospital at Herlev; Maria Wilcke, M.D., Ph.D., Principal Investigator — Karolinska Institutet; Turkka Anttila, M.D., Principal Investigator — Helsinki University Central Hospital; Annele Pönkkö, M.D., Principal Investigator — Oulu University Hospital; Jerzy Stiasny, M.D., Principal Investigator — Hospital Sønderjylland; Tuukka Tanskanen, M.D., Principal Investigator — Turku University Hospital
Locations (9):
- Denmark (2):
  - Herlev/Gentofte University Hospital of Copenhagen, Copenhagen
  - Hospital Sønderjylland, Sønderborg
- Finland (6):
  - Hospital Nova of Central Finland, Jyväskylä, Central Finland
  - Oulu University Hospital, Oulu, North Ostrobothnia
  - Kuopio University Hospital, Kuopio, Northern Savonia
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University Hospital, Helsinki, Uusimaa
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All the IPD will be shared with other researchers by request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after the publication and it will be available for 15 years.
Access Criteria: By request.

REFERENCES:
- [Derived] Kaivorinne A, Raisanen MP, Karjalainen T, Jokihaara J, Gvozdenovic R, Wilcke M, Reito A, Anttila T, Ponkko A, Lauridsen C, Tanskanen T, Mattila VM; REINFORCER investigators. tREatment of trIaNgular FibrOcaRtilage ComplEx Ruptures (REINFORCER): protocol for randomised, controlled, blinded, efficacy trial of triangular fibrocartilage complex tears. BMJ Open. 2024 Dec 11;14(12):e086102. doi: 10.1136/bmjopen-2024-086102. PMID 39663172